CLINICAL TRIAL: NCT06792136
Title: A Phase IIa, Randomized, Double-blind, Placebo Controlled, Parallel Group, Multi-center Trial to Evaluate the Efficacy and Safety of ONO-1110 in Patients With Major Depressive Disorder
Brief Title: A Study of ONO-1110 in Patients With Major Depressive Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-1110-07; jRCT2031240577 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder (MDD
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-1110 (Experimental)
  Interventions: Drug: ONO-1110; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: ONO-1110; Drug: Placebo

INTERVENTIONS:
Drug: ONO-1110 — ONO-1110 tablets once a day
Drug: Placebo — Placebo tablets once daily

SUMMARY:
To Evaluate the Efficacy and Safety of ONO-1110 in Patients with Major Depressive Disorder

ELIGIBILITY:
Inclusion Criteria:

1. Japanese (sex not specified)
2. Participants who, in the opinion of the principal (or sub-investigator), are capable of understanding the content of the clinical trial and complying with its requirements
3. Participants diagnosed with major depressive disorder based on DSM-5-TR (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision) criteria, as determined through an interview using the M.I.N.I. (Mini-international neuropsychiatric interview)
4. Outpatients
5. Participants whose current depressive episode has lasted for at least 2 months but no more than 12 months
6. Participants with a HAM-D17 (Hamilton depression rating scale 17 items) total score of 18 or higher and a CGI-S (Clinical global impression-Improvement) score of 4 or higher

Exclusion Criteria:

1. Participants with a current or past history of psychiatric or neurological disorders that meet any of the following criteria:

   * Participants with a comorbid psychiatric disorder other than major depressive disorder as defined by DSM-5-TR (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision) (assessed using the M.I.N.I.(Mini-international neuropsychiatric interview))
   * Participants with major depressive disorder with mixed features, psychotic features, or catatonia as defined by DSM-5-TR (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision)
   * Participants with a current or past history of schizophrenia or other psychotic disorders as defined by DSM-5-TR (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision)
   * Participants with neurodevelopmental disorders or personality disorders as defined by DSM-5-TR (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision)
   * Participants with a current or past history of clinically significant neurological disorders (including epilepsy)
   * Participants with neurodegenerative diseases (such as Alzheimer's disease, Parkinson's disease, multiple sclerosis, etc.)
2. Participants who, in the opinion of the principal (or sub-investigator), have not responded to at least two different antidepressants, each administered at an adequate dose for at least 6 weeks, during the current or past depressive episode.
3. Participants who have used adjunctive treatments such as lithium, triiodothyronine/thyroxine, lamotrigine, valproate, carbamazepine, or atypical antipsychotics, or who have used combination therapy with antidepressants for the current depressive episode.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in HAM-D17(Hamilton depression rating scale 17 items) total score from baseline to Week 8 of the treatment period | Up to 16 weeks

SECONDARY OUTCOMES:
The transition of HAM-D17(Hamilton depression rating scale 17 items) total score from baseline to Week 8 of the treatment period | Up to 16 weeks
Responder rates of HAM-D17(Hamilton depression rating scale 17 items) total score at 1, 2, 4, 6, and 8 weeks of the treatment period | Up to 16 weeks
  Responder is defined as a reduction of 50% or more in HAM-D17(Hamilton depression rating scale 17 items) total score from baseline
Remitted patient rates of HAM-D17(Hamilton depression rating scale 17 items) score at 1, 2, 4, 6, and 8 weeks of the treatment period | Up to 16 weeks
  Remitted patient is defined as a total HAM-D17(Hamilton depression rating scale 17 items) total score of 7 or less.
Change in the total MADRS(Montgomery-Åsberg depression rating scale) score from baseline to Week 8 of the treatment period | Up to 16 weeks
Transition of HAM-A(Hamilton Anxiety Scale) total score from baseline to Week 8 of the treatment period | Up to 16 weeks
Transition of CGI-S(Clinical Global Impression of illness Severity) score from baseline to Week 8 of the treatment period | Up to 16 weeks
Transition of QIDS-J(Quick Inventory of Depressive Symptomatology) total score from baseline to Week 8 of the treatment period | Up to 16 weeks
Transition of CGI-I(Clinical Global Impression of Impression Important) score from baseline to Week 8 of the treatment period | Up to 16 weeks
Plasma ONO-1110 concentrations | Up to 16 weeks
Adverse Events | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (29):
- Japan (29):
  - AK Clinic, Fukuoka
  - Hiro Mental Clinic, Fukuoka
  - Hirota Clinic, Fukuoka
  - Kokorono Clinic Hirao, Fukuoka
  - Kokorono Clinic Iizuka, Fukuoka
  - Kokura Mental Clinic, Fukuoka
  - Mental Clinic Sakurazaka, Fukuoka
  - Shinseikai Kaku Mental Clinic, Fukuoka
  - Uematsu Mental Clinic, Fukuoka
  - Ichikawa Clinic, Gunma
  - Higashi-Sapporo Mental Clinic, Hokkaido
  - Kawamura Mental Clinic, Hokkaido
  - Minami1jo Mental Clinic, Hokkaido
  - Sapporo Kobushi Clinic, Hokkaido
  - Shimode Mental Clinic, Hokkaido
  - Tatsuta Clinic, Hyōgo
  - Kishiro Mental Clinic, Kanagawa
  - Yutaka Clinic, Kanagawa
  - Harai Clinic, Tokyo
  - Iidabashi Mental Clinic, Tokyo
  - Ikebukuro Olive Mental Clinic, Tokyo
  - Kitaikebukuro Kokoro No Clinic, Tokyo
  - Maynds Tower Mental Clinic, Tokyo
  - Meguroeki Higashiguchi Mental Clinic, Tokyo
  - Monzen-nakacho Mental Clinic, Tokyo
  - Niseikai Murakami Iin, Tokyo
  - Nishi-Shinjuku Concieria Clinic, Tokyo
  - Sakurazaka Clinic SophyAnce, Tokyo
  - Sangenjaya Nakamura Mental Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: No